CLINICAL TRIAL: NCT07276295
Title: Synthetic Versus Autologous Sling For Stress Incontinence (SASSI): A Randomized Controlled Trial
Brief Title: Synthetic Versus Autologous Sling For Stress Incontinence
Acronym: SASSI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Roxana Geoffrion, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H25-02899
Record Dates: First submitted 2025-11-26; First posted 2025-12-11 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Urinary Incontinence
Keywords: autologous fascia sling; stress predominant urinary incontinence; tension-free vaginal tape
MeSH Terms: conditions — Urinary Incontinence | interventions — Suburethral Slings

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tension-free vaginal tape (Active Comparator)
  Interventions: Procedure: tension-free vaginal tape
- autologous fascia sling (Active Comparator)
  Interventions: Procedure: autologous fascia sling

INTERVENTIONS:
Procedure: autologous fascia sling — Participants will receive autologous fascia sling as surgery for stress predominant urinary incontinence.
  Arms: autologous fascia sling
Procedure: tension-free vaginal tape — Participants will receive tension-free vaginal tape as surgery for stress predominant urinary incontinence.
  Arms: tension-free vaginal tape

SUMMARY:
This is a multi-centre randomized controlled trial comparing mid-urethral synthetic mesh sling or tension-free vaginal tape (TVT) and autologous fascia sling (AFS) in elderly patients with stress predominant urinary incontinence. The investigators aim to investigate new onset pelvic pain 6 months post-op and objective urinary incontinence cure rate 5 years post-op. Secondary objectives include investigation of opioid use, mental health, sexual health, and other post-op outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult females at birth (female anatomy, any gender)
* Greater than or equal to 60 years old
* Have stress predominant urinary incontinence (spUI) eligible for both types of surgery (tension-free vaginal tape and autologous fascia sling)
* Exhausted conservative management options for UI (Kegel's exercises, physiotherapy, pessary)
* Completed childbearing
* Able to follow up with clinic visits for up to five years after surgery

Exclusion Criteria:

* Clinical Frailty Score of 6 or more, as moderate frailty is likely associated with excessive postoperative deterioration
* Concurrent pelvic surgery
* Neurogenic bladder
* Previous UI surgery
* Previous pelvic radiation
* Previous mesh exposure
* Presence of pelvic pain for more than three months in the last five years
* Likely unable to follow up
* Immunocompromised individuals receiving immunosuppressive medications for at least 3 months
* Chronic systemic steroid use for at least 3 months for autoimmune diseases
* Unable to stop smoking for at least 3 months prior to surgery and at high risk of restart smoking post-operatively

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2032-06 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Objective urinary incontinence status measured by standing cough test | 5 years post-op
  Unit of measure: proportion of participants Measurement tool: standing cough test positive, yes/no
Incidence of new-onset chronic abdominopelvic pain since surgery by Likert pain intensity scale | 6 months post-op
  Proportion of participants who report new abdominopelvic pain with an average intensity greater than 3 on a 0-10 Likert pain intensity scale over the past 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada